CLINICAL TRIAL: NCT03275896
Title: Evaluation of the Efficacy of Descemet Membrane Transplantation for the Treatment of Fuchs' Endothelial Dystrophy
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Singapore National Eye Centre (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: R1366/52/2016
Record Dates: First submitted 2017-09-04; First posted 2017-09-08 (Actual); Last update posted 2017-09-08 (Actual); Status verified 2017-09

CONDITIONS: Fuchs' Endothelial Dystrophy
MeSH Terms: conditions — Fuchs' Endothelial Dystrophy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Descemet Membrane Transplantation (Experimental): Patients with severe, symptomatic Fuch's Endothelial Dystrophy (FED) will be offered Descemet Membrane Transplantation (DMT) for their condition.
  Interventions: Other: Descemet Membrane Transplantation

INTERVENTIONS:
Other: Descemet Membrane Transplantation — The diseased host Descemet membrane will first be stripped, as per a standard Descemet Stripping Automated Endothelial Keratoplasty surgery. A cadaveric, acellular Descemet membrane graft will then be harvested and transplanted onto the host.

SUMMARY:
Fuchs Endothelial Dystrophy (FED) is a degenerative disease affecting the corneal endothelium. The current gold-standard for treatment of severe FED is endothelial keratoplasty, wherein a cadaveric Descemet's membrane / endothelium graft is transplanted. In this study, the investigators hypothesized that the transplantation of an acellular Descemet's membrane (i.e. Descemet Membrane Transplantation, 'DMT') may be equally efficacious in promoting recovery of endothelial function in this group of patients.

DETAILED DESCRIPTION:
Fuchs Endothelial Dystrophy (FED) is a degenerative disease affecting the corneal endothelium, characterized clinically by guttate excrescences on the posterior corneal surface and dysfunctional corneal endothelial cells. While patients are commonly asymptomatic in their early stages, advanced FED can be associated with significant corneal edema, scarring and impairment of visual function.

Patients with mild FED are usually managed conservatively with the application of topical hypertonic saline eyedrops. For patients with advanced FED, endothelial keratoplasty may often be necessary. In 2014, FED represented the most common indication for endothelial keratoplasty in the United States, accounting for 47.7% (13,817 cases) of all endothelial keratoplasty procedures performed nationwide. In Singapore, FED was the second most common indication for corneal transplantation.

Endothelial keratoplasty is associated with endothelial cell attrition in the range of 29.7% - 47% by the 3rd post-operative year. Additionally, the global demand for corneal graft material currently still far outstrips supply, critically limiting the number of patients who can potentially benefit from these surgical interventions. As such, there is a need explore alternative, sustainable strategies for the management of FED.

In 2009, Shah et al. reported the treatment of a 34 years old patient, with the combined pathologies of FED and Posterior Polymorphous Corneal Dystrophy (PPMD), by primary stripping of the central 4-5mm of Descemet's membrane without corneal graft transplantation ('Primary Descemetorhexis'). Contrary to conventional expectations, there was complete repopulation of the posterior corneal surface by corneal endothelial cells following the surgery, with best-corrected-visual-acuity (BCVA) of 6/7.5 achieved by the 6th post-operative month. In 2014, Moloney et al. published a similar report of a 54 years old patient, diagnosed with FED, successfully treated by Primary Descemetorhexis. Rapid endothelial recovery, as evidenced by a central endothelial cell count of 620 cells/mm2 and BCVA of 6/6, was achieved by approximately 6 weeks after the surgery. The success of these cases raised the prospect of Primary Descemetorhexis as a feasible alternative for the treatment of FED.

To gain a better understanding of the factors which may affect endothelial recovery following Primary Descemetorhexis, investigators performed an ex vivo human corneal endothelial cell culture experiment in which Primary Descemetorhexis was performed on cadaveric human cornea buttons, followed by ex vivo culture for a duration of 2 weeks to allow for endothelial recovery. A less invasive approach of denuding endothelial cells from the Descemet's membrane (DM), while maintaining anatomical integrity of the DM, was also assessed. The investigators found that advanced patient age and the absence of DM were significantly associated with slower endothelial recovery.

As such, the investigators hypothesized that the outcomes of Primary Descemetorhexis for the treatment of FED may be improved by DM transplantation following Primary Descemetorhexis ('DM Transplantation'). The main difference between the proposed technique of DM transplantation and conventional endothelial keratoplasty is that the DM transplant does not require the presence of a functional corneal endothelial monolayer on the graft. If successful, the greatest advantage of this approach would be to greatly expand the pool of donors who are eligible to provide cadaveric corneal graft tissue for transplantation.

ELIGIBILITY:
Inclusion Criteria:

1. Fuchs' Endothelial Dystrophy (FED) as defined by any of the following criteria:

   1. FED of at least Grade 4 on the Krachmer grading scale (i.e. greater than 5mm of confluent central corneal guttata)
   2. Best-corrected-visual-acuity of less than 6/12 in a patient clinically diagnosed with FED of any grade, in which poor visual acuity cannot be accounted by any other significant ophthalmic disease (e.g. cataracts, age-related macular degeneration, glaucoma, optic neuropathies)
2. Patients in the range of <85 years old will be recruited for this study
3. Only individuals with the mental capacity to provide informed consent will be included.
4. Patients who are willing and able to sign a written Informed Consent Form prior to any study-specific procedures will be included
5. Patients who are willing and able to return for scheduled follow-up examinations for up to 12 months after the surgery will be included

Exclusion Criteria:

Subjects that meet any of the following criteria will be excluded from participation:

1. Eyes which have previously been subject to any form of keratoplasty
2. An only-functioning eye in a patient who has lost visual potential in the contralateral eye
3. Patients with chronic, advanced FED who meet the above mentioned inclusion criteria, but whose disease is associated with significant stromal scarring to such an extent that will predictably impair post-operative visual recovery after DSAEK or DM transplant
4. Patients whose corneal endothelial disease may possibly be attributed to pathologies other than FED, including but not limited to pseudophakic bullous keratopathy, laser-peripheral-iridotomy induced bullous keratopathy, iridocorneal endothelial syndrome, Axenfeld Rieger syndrome, congenital hereditary endothelial dystrophy and any other anterior segment developmental anomalies
5. Patients with visually significant cataracts
6. Patients with diagnosed with visually significant retinal disease, including but not limited to age-related macular degeneration, myopic macular degeneration, diabetic retinopathy, diabetes related maculopathy, retinal vein occlusion related maculpathy, retinal dystrophies and previous retinal detachments.
7. Patients with any form of glaucoma
8. Patients diagnosed with visually significant, non-glaucomatous optic neuropathies, including but not limited to those related to ischemic (both arteritic and non-arteritic), toxic, nutritional, myopic, compression, infective and inflammatory causes
9. Patients who are pregnant, lactating, of child-bearing potential and not practising a medically approved method of birth control, or planning to become pregnant during the course of the trial, and patients with other conditions associated with fluctuation of hormones that could lead to refractive changes.

Ages: 21 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2016-09 (Actual); Primary Completion 2020-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Central Endothelial Cell Density | Measured monthly, for the first 6 post-operative months
  Central endothelial cell density will be determined using a specular microscope (Konan Medical), measured as number of cells per square millimetre, using the automated cell counting algorithm.

SECONDARY OUTCOMES:
Visual acuity | Measured monthly, for the first 6 post-operative months
  The visual acuity will be measured using the Snellen visual acuity scale, performed in a standardized room using a 6-metre visual acuity lane, by a fully qualified optometrist.

CONTACTS AND LOCATIONS:
Overall Officials: Jodhbir Mehta, FRCS, Principal Investigator — Singapore National Eye Centre
Locations (1):
- Singapore National Eye Centre, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No
No sharing of OPD with other researchers

REFERENCES:
- [Background] Soh YQ, Peh G, George BL, Seah XY, Primalani NK, Adnan K, Mehta JS. Predicative Factors for Corneal Endothelial Cell Migration. Invest Ophthalmol Vis Sci. 2016 Feb;57(2):338-48. doi: 10.1167/iovs.15-18300. PMID 26842752
- [Background] Arbelaez JG, Price MO, Price FW Jr. Long-term follow-up and complications of stripping descemet membrane without placement of graft in eyes with Fuchs endothelial dystrophy. Cornea. 2014 Dec;33(12):1295-9. doi: 10.1097/ICO.0000000000000270. PMID 25299425
- [Background] Bleyen I, Saelens IE, van Dooren BT, van Rij G. Spontaneous corneal clearing after Descemet's stripping. Ophthalmology. 2013 Jan;120(1):215. doi: 10.1016/j.ophtha.2012.08.037. No abstract available. PMID 23283191
- [Background] Moloney G, Chan UT, Hamilton A, Zahidin AM, Grigg JR, Devasahayam RN. Descemetorhexis for Fuchs' dystrophy. Can J Ophthalmol. 2015 Feb;50(1):68-72. doi: 10.1016/j.jcjo.2014.10.014. Epub 2014 Oct 31. PMID 25677286
- [Background] Shah RD, Randleman JB, Grossniklaus HE. Spontaneous corneal clearing after Descemet's stripping without endothelial replacement. Ophthalmology. 2012 Feb;119(2):256-60. doi: 10.1016/j.ophtha.2011.07.032. Epub 2011 Oct 7. PMID 21982414
- [Background] Kitagawa K, Kojima M, Sasaki H, Shui YB, Chew SJ, Cheng HM, Ono M, Morikawa Y, Sasaki K. Prevalence of primary cornea guttata and morphology of corneal endothelium in aging Japanese and Singaporean subjects. Ophthalmic Res. 2002 May-Jun;34(3):135-8. doi: 10.1159/000063656. PMID 12097795
- [Derived] Soh YQ, Poh SSJ, Peh GSL, Mehta JS. New Therapies for Corneal Endothelial Diseases: 2020 and Beyond. Cornea. 2021 Nov 1;40(11):1365-1373. doi: 10.1097/ICO.0000000000002687. PMID 34633355

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2017-08-28): https://cdn.clinicaltrials.gov/large-docs/96/NCT03275896/Prot_SAP_000.pdf
  • Informed Consent Form (2016-06-27): https://cdn.clinicaltrials.gov/large-docs/96/NCT03275896/ICF_001.pdf